CLINICAL TRIAL: NCT06924658
Title: the Impact of Metformin Use on Clinical Outcomes in Gouty Patients
Brief Title: Metformin in Safety and Efficacy in Gouty Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8746
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): this group will receive placebo in addition to the traditional lines of treatment of gout.
  Interventions: Other: placebo
- Metformin group (Active Comparator): This group will receive metformin (1000mg/day) in addition to the traditional lines of treatment of gout.
  Interventions: Drug: Metformin

INTERVENTIONS:
Other: placebo — Placebo will have the same look of metformin
  Arms: Control group
Drug: Metformin — Metformin, a biguanide, is used to manage diabetes by reducing insulin resistance and preventing comorbidities such as cerebrovascular and coronary artery disease, as well as providing renal protection to diabetic nephropathy patients
  Arms: Metformin group

SUMMARY:
The most frequent crystal arthropathy is gout, which is also the most prevalent cause of inflammatory arthritis. Gouty Patients frequently have excruciating pain and swelling in their joints. Gout is linked to decreased health-related quality of life and functional disability. Gout and its associated diseases have been shown to have a significant impact on patients mortality and morbidities. Metformin, a biguanide, is used to manage diabetes by reducing insulin resistance and preventing comorbidities such as cerebrovascular and coronary artery disease, as well as providing renal protection to diabetic nephropathy patients

ELIGIBILITY:
Inclusion Criteria:

* Gouty patients clinically diagnosed as gouty arthritis based on the American College of Rheumatology/European League Against Rheumatism criteria of gout.

Exclusion Criteria:

* Systemic disorders such as cardiovascular, neurological, coronary artery disease.
* Hypertension, hyperlipidemia, diabetes mellitus, active infections.
* Other inflammatory or autoimmune diseases.
* Patients on biologics,
* Cases with hypersensitivity to metformin and those with impaired liver and kidney functions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
- Clinical assessment of disease activity | 3 months
  - Clinical assessment of disease activity by assessing patient and physician VAS visual analog scale (0-10 cm);

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt